CLINICAL TRIAL: NCT03524118
Title: A Double-blind, Randomized, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MK-1654 in Pre-Term and Full-Term Infants
Brief Title: Safety, Tolerability, and Pharmacokinetics of Clesrovimab (MK-1654) in Infants (MK-1654-002)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 1654-002; MK-1654-002 (Other: Merck Protocol Number); 2017-005062-21 (EudraCT Number)
Record Dates: First submitted 2018-05-11; First posted 2018-05-14 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Tract Infection; Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Tract Infections | interventions — MK-1654

STUDY DESIGN:
Intervention Model Description: Single ascending dose
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Panel A: Pre-term clesrovimab Dose 1 (Experimental): Pre-term infants will receive clesrovimab Dose 1 via intramuscular (IM) injection and will be followed for up to 365 days.
  Interventions: Drug: Clesrovimab
- Panel B: Pre-term clesrovimab Dose 2 (Experimental): Pre-term infants will receive clesrovimab Dose 2 via IM injection and will be followed for up to 365 days.
  Interventions: Drug: Clesrovimab
- Panel C: Pre-term clesrovimab Dose 3 (Experimental): Pre-term infants will receive clesrovimab Dose 3 via IM injection and will be followed for up to 365 days.
  Interventions: Drug: Clesrovimab
- Panel D1: Pre-term clesrovimab Dose 4 (Experimental): Pre-term infants enrolled prior to AM4 will receive clesrovimab Dose 4 via IM injection and will be followed for up to 365 days.
  Interventions: Drug: Clesrovimab
- Panel D2: Pre-term clesrovimab Dose 4 (Experimental): Pre-term infants enrolled after AM4 will receive clesrovimab Dose 4 via IM injection and will be followed for up to 545 days.
  Interventions: Drug: Clesrovimab
- Panel E1: Full-term clesrovimab Dose 4 (Experimental): Full-term infants enrolled prior to AM4 will receive clesrovimab Dose 4 via IM injection and will be followed for up to 365 days.
  Interventions: Drug: Clesrovimab
- Panel E2: Full-term clesrovimab Dose 4 (Experimental): Full-term infants enrolled after AM4 will receive clesrovimab Dose 4 via IM injection and will be followed for up to 545 days.
  Interventions: Drug: Clesrovimab
- Placebo (Placebo Comparator): Pre-term infants will receive placebo via IM injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clesrovimab — Single ascending doses of clesrovimab will be administered via IM injection.
  Other Names: MK-1654
  Arms: Panel A: Pre-term clesrovimab Dose 1; Panel B: Pre-term clesrovimab Dose 2; Panel C: Pre-term clesrovimab Dose 3; Panel D1: Pre-term clesrovimab Dose 4; Panel D2: Pre-term clesrovimab Dose 4; Panel E1: Full-term clesrovimab Dose 4; Panel E2: Full-term clesrovimab Dose 4
Drug: Placebo — Placebo (0.9% sodium chloride [NaCl]) will be administered via IM injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and incidence of anti-drug antibodies (ADAs) of single ascending doses of clesrovimab in healthy pre-term (born at 29 to 35 weeks gestational age) and full-term (born at >35 weeks gestational age) infants. Participants will be randomized into 1 of 4 dose escalation panels (Panels A to D); an additional panel (Panel E) of full-term infants will receive the same dose as Panel D. Key safety and tolerability variables will be reviewed after each dose panel prior to administering the next-highest dose.

DETAILED DESCRIPTION:
Participants in Dose Panels A, B, C, D1, and E1 will be followed for up to 365 days. After protocol Amendment 4 (AM4), participants in Dose Panels D2 and E2 will be followed for up to 545 days.

ELIGIBILITY:
Inclusion Criteria:

* is healthy, based on screening safety laboratory, medical history, and physical examination results
* is a pre-term infant (born at 29 weeks to 35 weeks gestational age [inclusive]) or a full-term infant (born at over 35 weeks gestational age), as confirmed in medical records
* weighs ≥2 kg at screening

Exclusion Criteria:

* has been recommended to receive palivizumab per local standard of care
* has ≥1 documented out-of-range safety laboratory results (adjusted for age) at the time of screening
* has a known hypersensitivity to any component of the respiratory syncytial virus (RSV) monoclonal antibody
* has a history of congenital or acquired immunodeficiency (e.g., splenomegaly)
* has documented human immunodeficiency virus (HIV) infection, hepatitis B (HBsAg positive), or hepatitis C (HCV ribonucleic acid [RNA] positive)
* has known history of functional or anatomic asplenia
* has a diagnosis of failure to thrive within 14 days of screening
* has known or history of a coagulation disorder contraindicating intramuscular injection
* has received or is expected to receive blood products (except irradiated platelets) within 3 months prior to enrollment
* has prior known documented RSV infection
* has hemodynamically significant congenital heart disease
* has chronic lung disease of prematurity requiring ongoing medical therapy
* has a history or current evidence of any condition, therapy, lab abnormality or other circumstance that, in the opinion of the investigator, might expose the participant to undue risk by participating in the study, confound the results of the study, or interfere with the participant's participation for the full duration of the study
* has any history of malignancy prior to randomization
* if any of the following apply, the Day 1 visit may be rescheduled for a time when these criteria are not met:
* has had a recent febrile illness (rectal temperature 38.1°C [100.5°F] or higher or axillary temperature 37.8°C [100.0°F] or higher) within 72 hours pre-dose
* is not up-to-date on required vaccinations per local pediatric vaccine schedule at time of screening
* has received inactivated or component vaccines (eg, influenza, hepatitis B) less than 14 days pre-dose
* has received live, attenuated, non-study licensed pediatric vaccines (e.g., Bacillus Calmette-Guerin vaccine) less than 30 days pre-dose
* has received any prior vaccine or monoclonal antibody (mAb) for the prevention of RSV
* is currently participating in or has participated in an interventional clinical study with an investigational compound or device at any time prior to first dose administration or while participating in this current study (participants enrolled in observational studies may be included and will be reviewed on a case-by-case basis for approval by the Sponsor)
* has enrolled previously in this study and been discontinued
* participant's mother participated in a RSV vaccine clinical study while pregnant and participant is ≤3 months of chronological age
* is unable to provide blood sample at screening
* cannot be adequately followed for safety according to the protocol plan
* has a parent/legally acceptable representative who is unlikely to adhere to study procedures, keep appointments, or is planning to relocate during the study
* is, or has, an immediate family member (eg, spouse, parent/guardian, sibling, or child) who is directly involved with the study at the site or with the Sponsor

Ages: 2 Weeks to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (34):
- United States (17):
  - Children's Hospital - Colorado ( Site 0067), Aurora, Colorado
  - Next Phase Research Alliance, LLC ( Site 0075), Homestead, Florida
  - Acevedo Clinical Research Associates ( Site 0025), Miami, Florida
  - Kapiolani Medical Center for Women and Children ( Site 0027), Honolulu, Hawaii
  - Cotton-O'Neil Clinical Research Center PediatricCare ( Site 0081), Topeka, Kansas
  - Children's Mercy Hospital ( Site 0037), Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center ( Site 0032), Lebanon, New Hampshire
  - SUNY Upstate Medical University Hospital ( Site 0029), Syracuse, New York
  - WakeMed Health and Hospitals ( Site 0033), Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center ( Site 0031), Cincinnati, Ohio
  - Ohio Pediatric Research Association ( Site 0066), Dayton, Ohio
  - Coastal Pediatric Research ( Site 0028), Charleston, South Carolina
  - Tribe Clinical Research, LLC ( Site 0082), Greenville, South Carolina
  - University of Texas Medical Branch at Galveston ( Site 0039), Galveston, Texas
  - Tekton Research, Inc. ( Site 0026), San Antonio, Texas
  - Multicare Institute For Research And Innovation ( Site 0035), Tacoma, Washington
  - University of Wisconsin American Family Children's Hospital ( Site 0068), Madison, Wisconsin
- Chile (4):
  - Centro de Investigacion Clinica Bradford Hill ( Site 0103), Santiago, Region M. de Santiago
  - Hospital La Florida ( Site 0050), Santiago, Region M. de Santiago
  - Facultad Medicina Universidad de Chile ( Site 0104), Santiago, Region M. de Santiago
  - Hospital Padre Hurtado ( Site 0102), Santiago, Region M. de Santiago
- Colombia (6):
  - Fundacion Hospital San Vicente de Paul ( Site 0097), Medellín, Antioquia
  - Universidad Pontificia Bolivariana - Clinica Universitaria Bolivariana ( Site 0098), Medellín, Antioquia
  - MedPlus Medicina Prepagada S.A. ( Site 0095), Bogotá, Bogota D.C.
  - Fundacion Universitaria de Ciencias de la Salud - Sociedad de Cirugia ( Site 0099), Bogotá, Bogota D.C.
  - Centro de Atención e Investigación Médica SAS - CAIMED CHIA ( Site 0100), Chía, Cundinamarca
  - Fundacion Valle del Lili ( Site 0090), Cali, Valle del Cauca Department
- South Africa (2):
  - Chris Hani Baragwanath Academic Hospital ( Site 0262), Johannesburg, Gauteng
  - Tygerberg Hospital ( Site 0261), Cape Town, Western Cape
- South Korea (3):
  - Seoul National University Hospital ( Site 0071), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0073), Seoul
  - Samsung Medical Center ( Site 0072), Seoul
- Spain (2):
  - Hospital Clinico Universitario de Santiago ( Site 0241), Santiago de Compostela, La Coruna
  - Hospital Universitario La Paz ( Site 0242), Madrid

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Madhi SA, Simoes EAF, Acevedo A, Novoa Pizarro JM, Shepard JS, Railkar RA, Cao X, Maas BM, Zang X, Krick A, Roadcap B, Vora KA, Aliprantis AO, Lee AW, Sinha A. A Phase 1b/2a Trial of a Half-life Extended Respiratory Syncytial Virus Neutralizing Antibody, Clesrovimab, in Healthy Preterm and Full-term Infants. J Infect Dis. 2025 Mar 17;231(3):e478-e487. doi: 10.1093/infdis/jiae581. PMID 39601265
- [Result] Thambi N, Phuah JY, Staupe RP, Tobias LM, Cao Y, McKelvey T, Railkar RA, Aliprantis AO, Arriola CS, Maas BM, Vora KA. Development of High-Titer Antidrug Antibodies in a Phase 1b/2a Infant Clesrovimab Trial Are Associated With RSV Exposure Beyond Day 150. J Infect Dis. 2025 Mar 17;231(3):e488-e496. doi: 10.1093/infdis/jiae582. PMID 39590882
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 183 participants were randomized and 181 were dosed and included in the All Participants as Treated (APaT) population. Two participants who were randomized to the MK-1654 20 mg dose group actually received MK-1654 50 mg and were included in the MK-1654 50 mg group for safety, pharmacokinetic (PK) and immunogenicity analyses.
Pre-assignment Details: Participants enrolled in panels D and E prior to protocol amendment 04 who chose not to participate in the modified schedule followed the D1 and E1 schedule of activities. Participants enrolled in panels D and E prior to protocol amendment 04 who chose to participate in the modified schedule followed the D2 and E2 schedule of activities.
Groups:
- Panel A: Preterm Clesrovimab 20mg: Pre-term infants received clesrovimab 20mg via intramuscular (IM) injection and were followed for up to 365 days.
- Panel B: Pre-term Clesrovimab 50mg: Pre-term infants received clesrovimab 50mg via IM injection and were followed for up to 365 days.
- Panel C: Pre-term Clesrovimab 75mg: Pre-term infants received clesrovimab 75mg via IM injection and were followed for up to 365 days.
- Panel D1 and D2: Pre-term Clesrovimab 100mg: Pre-term infants in Panel D1 and D2 received clesrovimab 100mg via IM injection and were followed for up to 365 and 545 days respectively.
- Panel E1 and E2: Full-term Clesrovimab 100mg: Full-term infants in Panel E1 and E2 received clesrovimab 100mg via IM injection and were followed for up to 365 and 545 days respectively.
- Placebo: Pre-term and Full-term infants received placebo via IM injection.
Period: Overall Study
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg | Placebo
Started | 8 | 31 | 41 | 32 | 33 | 38
Treated | 8 | 31 | 40 | 32 | 32 | 38
Safety Analysis Population (Two participants who were randomized to the MK-1654 20 mg dose group actually received MK-1654 50 mg) | 6 | 33 | 40 | 32 | 32 | 38
Completed | 8 | 29 | 40 | 31 | 26 | 37
Not Completed | 0 | 2 | 1 | 1 | 7 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 1 | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panel D1 and D2: Pre-term Clesrovimab 100mg: Pre-term infants received clesrovimab 100mg via IM injection and were followed for up to 365 and 545 days.
- Panel E1 and E2: Full-term Clesrovimab 100mg: Full-term infants received clesrovimab 100mg via IM injection and were followed for up to 365 and 545 days.
- Total: Total of all reporting groups
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg | Placebo | Total
Number analyzed (Participants) | 8 | 31 | 41 | 32 | 33 | 38 | 183
Age, Continuous [Median (Full Range); unit: days] | 68.0 [31 to 257] | 109.0 [23 to 255] | 94.0 [24 to 245] | 139.5 [14 to 239] | 164.0 [46 to 250] | 128.0 [26 to 275] | 126.0 [14.0 to 275]
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 2 | 3 | 3 | 0 | 2 | 10
  Infants and toddlers (28 days-23 months) | 8 | 29 | 38 | 29 | 33 | 36 | 173
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 20 | 17 | 13 | 19 | 90
  Male | 2 | 16 | 21 | 15 | 20 | 19 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 12 | 25 | 9 | 14 | 18 | 79
  Not Hispanic or Latino | 7 | 19 | 16 | 23 | 19 | 20 | 104
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 1 | 2 | 5
  Asian | 0 | 1 | 0 | 5 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 8 | 9 | 14 | 14 | 11 | 60
  White | 4 | 20 | 14 | 8 | 11 | 14 | 71
  More than one race | 0 | 1 | 17 | 2 | 7 | 9 | 36
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced At Least One Solicited Injection Site Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection site AEs were monitored from Day 1 to Day 5.
Time Frame: Up to Day 5
Population: Safety analysis population consisted of all participants who received at least one dose of study treatment. Two participants who were randomized to the MK-1654 Panel A 20 mg dose group actually received MK-1654 Panel B 50mg and were included in the MK-1654 50 mg group for the protocol specified safety analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg | Placebo
Number analyzed (Participants) | 6 | 33 | 40 | 32 | 32 | 38
Participants
  with solicited injection site adverse events | 3 | 3 | 3 | 2 | 2 | 2
  without solicited injection site adverse events | 3 | 30 | 37 | 30 | 30 | 36

2. Primary Outcome: Percentage of Participants Who Experienced At Least One Solicited Systemic Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs were monitored from Day 1 to Day 5.
Time Frame: Up to Day 5
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg | Placebo
Number analyzed (Participants) | 6 | 33 | 40 | 32 | 32 | 38
Participants
  with solicited systemic adverse events | 2 | 8 | 9 | 2 | 3 | 9
  without solicited systemic adverse events | 4 | 25 | 31 | 30 | 29 | 29

3. Primary Outcome: Percentage of Participants Who Experienced At Least One Serious Adverse Event (SAE)
Description: An SAE is any untoward medical occurrence that, at any dose, results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant injury/incapacity; is a congenital anomaly/birth defect; or is an other important medical event.
Time Frame: Up to Day 545
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg | Placebo
Number analyzed (Participants) | 6 | 33 | 40 | 32 | 32 | 38
Participants
  with serious adverse events (SAE) | 1 | 4 | 1 | 3 | 6 | 6
  without SAE | 5 | 29 | 39 | 29 | 26 | 32

4. Secondary Outcome: Area Under the Serum-Concentration Time Curve From Zero to Infinity (AUC0-∞)
Description: AUC0-∞ is a measure of the extrapolated mean concentration in serum from dosing to infinity.
Time Frame: At designated time points (up to 1 year post-dose)
Population: All randomized participants who received at least one dose of study treatment, with exclusions for important protocol deviations that may have substantially affected the results and with data available for this outcome measure. Two participants who were randomized to the MK-1654 Panel A 20 mg dose group actually received MK-1654 Panel B 50mg and were included in the MK-1654 50 mg group for the protocol specified PK analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
day*μg/mL | 1560 (43.5) | 3520 (22.8) | 5510 (22.4) | 6790 (25.4) | 5690 (15.9)

5. Secondary Outcome: Maximum Serum Concentration (Cmax) of Clesrovimab
Description: Cmax is the highest observed serum drug concentration.
Time Frame: At designated time points (up to 1 year post-dose)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
μg/mL | 26.3 (19.3) | 61.7 (21.8) | 94.5 (20.5) | 117 (23.5) | 99.9 (13.7)

6. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Clesrovimab
Description: Tmax is the time taken to reach the maximum observed plasma (Cmax) concentration of Clesrovimab.
Time Frame: At designated time points (up to 1 year post-dose)
Population: as for outcome 4
Measure: Median (Full Range); unit: day
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
day | 4.0 [3.8 to 4.60] | 4.20 [3.70 to 5.30] | 4.20 [3.00 to 5.80] | 4.10 [3.70 to 6.00] | 4.10 [3.70 to 4.90]

7. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Clesrovimab
Description: t1/2 is the time required for 50% of drug to be cleared from serum.
Time Frame: At designated time points (up to 1 year post-dose)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
day | 48.8 (34.6) | 44.6 (10.9) | 46.1 (15.1) | 45.2 (13.7) | 43.0 (9.72)

8. Secondary Outcome: Serum Concentration of Clesrovimab on Day 7 (C7days)
Description: Serum concentration of clesrovimab was measured on Day 7.
Time Frame: Day 7
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
μg/mL | 24.4 (20.4) | 57.8 (21.6) | 88.1 (20.4) | 109 (23.0) | 92.8 (13.3)

9. Secondary Outcome: Serum Concentration of Clesrovimab on Day 14 (C14days)
Description: Serum concentration of clesrovimab was measured on Day 14.
Time Frame: Day 14
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
μg/mL | 19.4 (22.1) | 46.8 (20.6) | 71.1 (19.7) | 88.6 (21.8) | 75.4 (12.9)

10. Secondary Outcome: Serum Concentration of Clesrovimab on Day 90 (C90days)
Description: Serum concentration of clesrovimab was measured on Day 90.
Time Frame: Day 90
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
μg/mL | 5.60 (49.5) | 13.0 (25.4) | 20.4 (25.8) | 25.2 (28.6) | 21.1 (18.8)

11. Secondary Outcome: Serum Concentration of Clesrovimab on Day 150 (C150days)
Description: Serum concentration of clesrovimab was measured on Day 150.
Time Frame: Day 150
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
μg/mL | 2.24 (80.6) | 4.98 (34.2) | 8.05 (37.7) | 9.70 (40.2) | 7.96 (26.7)

12. Secondary Outcome: Serum Concentration of Clesrovimab on Day 365 (C365days)
Description: Serum concentration of clesrovimab was measured on Day 365.
Time Frame: Day 365
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 5 | 33 | 40 | 32 | 31
μg/mL | 0.0953 (362) | 0.177 (79.4) | 0.313 (107) | 0.355 (104) | 0.248 (63.1)

13. Secondary Outcome: Number of Participants With Positive Titer of Anti-Drug Antibodies (ADAs) for Clesrovimab: Panels A, B, C, D1, D2, E1, and E2
Description: ADA was assessed at 2 or 3 of the following timepoints for each participant: Days 14, 90, 150, 365 and 545. ADA status for each participant was determined across the timepoints assessed. The definitions of the categories are as follows: (1) ADA Negative: participants whose ADA results were negative at all timepoints measured; (2) Non-treatment emergent positive: participants whose ADA result was positive only at baseline or if postdose titer increased by less than 2-fold relative to the baseline titer; (3) Positive response to MK-1654: participants whose ADA result was negative at baseline and positive at one or more postdose timepoints or participants whose ADA result was positive at baseline and postdose titer increased by greater than or equal to 2-fold relative to the baseline titer.
Time Frame: Days 14, 90, 150, 365 and 545
Population: All randomized participants who received at least one dose of study treatment and were evaluable with at least one ADA result after treatment with MK-1654. Two participants who were randomized to the MK-1654 Panel A 20 mg dose group actually received MK-1654 Panel B 50 mg and were included in the MK-1654 50 mg group for the protocol specified immunogenicity analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Preterm Clesrovimab 20mg | Panel B: Pre-term Clesrovimab 50mg | Panel C: Pre-term Clesrovimab 75mg | Panel D1 and D2: Pre-term Clesrovimab 100mg | Panel E1 and E2: Full-term Clesrovimab 100mg
Number analyzed (Participants) | 6 | 32 | 39 | 32 | 30
Participants
  ADA Negative status | 4 | 23 | 35 | 15 | 9
  Non-treatment emergent positive | 0 | 0 | 0 | 1 | 1
  ADA Positive response to MK-1654 | 2 | 9 | 4 | 16 | 20
  Maximum Postdose Titer of 20 to < 189 of ADA | 0 | 6 | 2 | 4 | 2
  Maximum Postdose Titer of 189 to < 1077.5 of ADA | 0 | 1 | 1 | 3 | 7
  Maximum Postdose Titer of 1077.5 to < 9285 of ADA | 0 | 0 | 1 | 4 | 7
  Maximum Postdose Titer of 9285 to 160000 of ADA | 2 | 2 | 0 | 4 | 4

ADVERSE EVENTS:
Time Frame: Up to Day 545
Description: All-cause mortality was analyzed in all randomized participants. AEs were analyzed in all participants who received at least one dose of study treatment. Additionally, two participants who were randomized to the MK-1654 Panel A 20 mg dose group actually received MK-1654 Panel B 50mg and were included in the MK-1654 50 mg group for the protocol specified safety analysis population.
Groups:
- MK-1654 20 mg in Pre-term Infants: Pre-term infants received clesrovimab 20mg via intramuscular (IM) injection and were followed for up to 365 days.
- MK-1654 50 mg in Pre-term Infants: Pre-term infants received clesrovimab 50mg via IM injection and were followed for up to 365 days.
- MK-1654 75 mg in Pre-term Infants: Pre-term infants received clesrovimab 75mg via IM injection and were followed for up to 365 days.
- MK-1654 100 mg Pre-Term Infants: Pre-term infants in Panel D1 and D2 received clesrovimab 100mg via IM injection and were followed for up to 365 and 545 days respectively.
- MK-1654 100 mg Full-Term Infants: Full-term infants in Panel E1 and E2 received clesrovimab 100mg via IM injection and were followed for up to 365 and 545 days respectively.
Arm/Group | MK-1654 20 mg in Pre-term Infants | MK-1654 50 mg in Pre-term Infants | MK-1654 75 mg in Pre-term Infants | MK-1654 100 mg Pre-Term Infants | MK-1654 100 mg Full-Term Infants | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/31 | 0/41 | 0/32 | 0/33 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/33 | 1/40 | 3/32 | 6/32 | 6/38
Other Adverse Events (participants affected / at risk) | 6/6 | 29/33 | 29/40 | 26/32 | 29/32 | 33/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1654 20 mg in Pre-term Infants (N=6) | MK-1654 50 mg in Pre-term Infants (N=33) | MK-1654 75 mg in Pre-term Infants (N=40) | MK-1654 100 mg Pre-Term Infants (N=32) | MK-1654 100 mg Full-Term Infants (N=32) | Placebo (N=38)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irregular breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1654 20 mg in Pre-term Infants (N=6) | MK-1654 50 mg in Pre-term Infants (N=33) | MK-1654 75 mg in Pre-term Infants (N=40) | MK-1654 100 mg Pre-Term Infants (N=32) | MK-1654 100 mg Full-Term Infants (N=32) | Placebo (N=38)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (2) | 2 (2) | 4 (4) | 5 (5)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (2)
Injection site swelling (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Bronchiolitis (Infections and infestations) | 2 (3) | 2 (3) | 4 (6) | 7 (8) | 5 (6) | 5 (9)
Bronchitis (Infections and infestations) | 0 (0) | 3 (7) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (8) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (7) | 11 (19) | 10 (20) | 10 (22) | 7 (19)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 3 (3)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 17 (22) | 7 (8) | 12 (19) | 18 (52) | 12 (22)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 5 (7)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 4 (4)
Irritability (Psychiatric disorders) | 2 (2) | 7 (7) | 5 (6) | 2 (2) | 2 (2) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 3 (8) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6) | 2 (2) | 6 (6) | 8 (11) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (6) | 3 (11) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03524118/Prot_SAP_000.pdf